CLINICAL TRIAL: NCT04771637
Title: Effect of Dexmedetomidine on Perioperative Internal Environment and Rehabilitation of Patients Undergoing Gastrointestinal Malignant Tumor Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20210213
Record Dates: First submitted 2021-02-13; First posted 2021-02-25 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-02

CONDITIONS: Dexmedetomidine; Perioperative; Electrolyte
Keywords: Dexmedetomidine; Electrolyte; Haemodynamics; Rehabilitation; Internal environment
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control with normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline
- dexmedetomidine loading dose 1 µg/kg + maintenance dose 0.25 µg/kg/h (Experimental)
  Interventions: Drug: Dexmedetomidine
- dexmedetomidine loading dose 0.5 µg/kg + maintenance dose 0.5 µg/kg/h (Experimental)
  Interventions: Drug: Dexmedetomidine
- dexmedetomidine loading dose 1 µg/kg + maintenance dose 0.5 µg/kg/h (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The loading dose with 0.5 μg/kg, maintenance dose with 0.5 μg/kg of Dexmedetomidine is used to observe the effect on the electrolyte and quality of recovery of the patients
  Arms: dexmedetomidine loading dose 1 µg/kg + maintenance dose 0.25 µg/kg/h
Drug: Dexmedetomidine — The loading dose with 1.0 μg/kg, maintenance dose with 0.25 μg/kg of Dexmedetomidine is used to observe the effect on the electrophysiology and quality of recovery of the patient
  Arms: dexmedetomidine loading dose 0.5 µg/kg + maintenance dose 0.5 µg/kg/h
Drug: Dexmedetomidine — The loading dose with 1 μg/kg, maintenance dose with 0.5 μg/kg of Dexmedetomidine is used to observe the effect on the electrophysiology and quality of recovery of the patients
  Arms: dexmedetomidine loading dose 1 µg/kg + maintenance dose 0.5 µg/kg/h
Drug: Normal saline — Normal saline is used to observe the effect on the electrophysiology and quality of recovery of the patients
  Arms: control with normal saline

SUMMARY:
Dexmedetomidine is a highly selective alpha2-adrenergic receptor agonist with sedative, analgesic, anti-anxiety, and inhibitory sympathetic nerve excitation properties. It is commonly used in clinical anesthesia and intensive care.Radical gastrectomy for gastrointestinal malignant tumors is a common major operation in clinical practice, with long operation time, great trauma and strong stress response of patients. Dexmedetomidine is often used in general anesthesia during such operations, but its long-term use or large dose may produce certain side effects.Common side effects of dexmedetomidine include bradycardia and hypotension, etc. Previous studies have reported that dexmedetomidine can prolong QT interval and is at risk of causing tip torsion type ventricular tachycardia.Abnormal Potassium may affect myocardial repolarization and increase the risk of tip torsion ventricular tachycardia.The main purpose of this study was to observe the effects of long-term use of dexmedetomidine on perioperative internal environment such as electrolyte and rehabilitation indicators during radical general anesthesia for gastrointestinal malignancy, and the secondary purpose was to explore the optimal dose of dexmedetomidine for general anesthesia for patients undergoing radical general anesthesia for gastrointestinal malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I or II;
2. age between 50-75 years, and a body mass index (BMI) between 18.5-28 kg/m2.

Exclusion Criteria:

1. Patients whoused hormones or drugs that have a hypoglycemic nature during the preoperative state, or had bradycardia, arrhythmia, hypotension, abnormal liver or kidney function, pancreatic disease, neuroendocrine malignancy, intraoperative blood transfusion;
2. Patients who refused participation and those who needed intensive care after the surgery were also excluded from the study;
3. Patients who had severe internal environmental disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
age | perioperative
  the age(years)
weight | perioperative
  weight(kg)
height | perioperative
  height(m)
sex | perioperative
  sex(male/female)
ASA status | perioperative
  ASA status of patients

SECONDARY OUTCOMES:
internal environment | Day 1
  the concentrations of sodium(mmol/L), lactate(mmol/L), potassium(mmol/L), calcium(mmol/L), base excess(mmol/L), base excess in the extracellular fluid compartment(mmol/L) were measured before the dexmedetomidine infusion (t1), 1 h after the surgery began (t2), at the end of the surgery (t3), and 1 h after transfer to the PACU (t4), 24h after the surgery

OTHER OUTCOMES:
drugs | 1 day
  the dosage of propofol, remifentanil and ephedrine
blood pressure | into PACU 30 minutes
  records the systolic blood pressure(mmHg), diastolic blood pressure(mmHg), and mean blood pressure(mmHg) of preoperative (T1), after infusion of loading dose of dexmedetomidine (T2), operation start (T3), operation start 5 min (T4), operation start 10 min (T5), operation start 1 h (T6), operation end(T7), immediately after extubation (T8), 5 min after extubation (T9) and into PACU 30 minutes (T10)
heart rate | into PACU 30 minutes
  records the heart rate(beats/minute) of preoperative (T1), after infusion of loading dose of dexmedetomidine (T2), operation start (T3), operation start 5 min (T4), operation start 10 min (T5), operation start 1 h (T6), operation end(T7), immediately after extubation (T8), 5 min after extubation (T9) and into PACU 30 minutes (T10)

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China